CLINICAL TRIAL: NCT00805844
Title: Monitoring Depth of Anesthesia With the SedLine Facilitates Motor Evoked Potential (MEP) Monitoring During Corrective Spinal Surgery
Brief Title: Motor Evoked Potentials and SedLine
Status: Terminated | Type: Observational
Why Stopped: Sponsor terminated the study
Sponsor: University of California, San Francisco (Other)
Responsible Party: Adrian W Gelb, Professor, UCSF
Other Study IDs: H50805-31889
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Spine Surgery
Keywords: Spine; Motor Evoked Potentials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Spine surgery with Motor Evoked Potential monitoring without SedLine monitoring visible.
- 2: Spine surgery with Motor Evoked Potential Monitoring with SedLine monitoring visible.

SUMMARY:
To determine if using usual clinical practice plus a depth of anesthesia monitor, SedLine, to guide anesthetic administration improves the quality and ease of MEP monitoring in patients undergoing corrective spinal procedures.

DETAILED DESCRIPTION:
Motor Evoked Potential (MEP) monitoring during spine surgery is now used routinely. However it is affected by a variety of anesthetics including fluctuating and/or excessively deep or light levels of anesthesia. A common problem is maintaining an overall constancy and adequacy of anesthesia. Individual patients' responses to anesthesia can differ greatly from population means and can complicate the interpretation of MEPs. False alarms can have significant consequences. One strategy to minimize the anesthetic induced variability of MEPs, and thereby improve the monitoring overall, is to keep the patient's anesthetic state (or "depth") in a narrow range during surgery. This study tests whether using a commercially available depth of anesthesia monitor in addition to usual clinical practice improves the quality of MEPs.

The hypothesis of this study is that the SedLine Monitor, which uses an EEG derived assessment of anesthetic depth, may facilitate MEP monitoring if it is kept within a narrow range during spine surgery. Because SedLine recommends maintaining their Index between 30 and 40 during surgical anesthesia, this is the range used in the primary hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing corrective spinal procedures, for whom MEP monitoring has been requested by the surgeon.
* 18 yrs of age or older

Exclusion Criteria:

* Minors, prisoners and those unable to consent for themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing corrective spinal procedures, for whom MEP monitoring has been requested by the surgeon.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is a composite measure of the motor evoked responses over the duration of the surgical procedure utilizing the "area under the curve" (AUC, volt-seconds) of the response time series | End of study

SECONDARY OUTCOMES:
Secondary outcomes include i) Stimulation threshold ii) MEP fade index and iii) Facilitation necessity and stability. | end of study

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States